CLINICAL TRIAL: NCT05176236
Title: Develop a Pictographic Educational Handouts and Validate Its Preliminary Efficacy on Tracheostomy Care
Brief Title: Pictographic Education Handout on Tracheostomy Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Sigma Theta Tau International Honor Society of Nursing (Other); University Hospitals Seidman Cancer Center (Other)
Responsible Party: Principal Investigator, Tongyao Wang, Research Fellow, Sarah Cole Hirsh Institute for Evidence Based Practice, Frances Payne Bolton School of Nursing, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pictograph_2021_STTI
Record Dates: First submitted 2021-10-13; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Health Literacy
Keywords: tracheostomy care; participatory action research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pictographic group (Experimental): Participants received the pictographic handouts on tracheostomy care
  Interventions: Other: Pictographic tracheostomy care handouts

INTERVENTIONS:
Other: Pictographic tracheostomy care handouts — The handouts were developed and validated by Clinical and inter-professional experts based on the hospital's text-based tracheostomy home care instructions.

SUMMARY:
The goal of the study is to address the clinical problem of poor education outcome from the current practice of teaching tracheostomy care by providing them with a pictographic education handout to assist their learning. The study seeks to establish face validity and preliminary efficacy of a pictographic education handout with patients and identify factors associated with lower self-efficacy level on tracheostomy care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Had a tracheostomy as part of head and neck cancer treatment, and who is not on mechanical ventilation
* His or her date of the related tracheostomy surgery was within the past 6 months
* Have received the discharge tracheostomy care education from the clinical nurse

Exclusion Criteria:

* Documented major physical or cognitive disabilities that would limit the ability to give informed consent or answer survey questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Author-developed self-efficacy on tracheostomy care scale | immediately after consenting and post intervention (up to 2 weeks) on study survey
  Participants' self-reported confidence on tracheostomy care from 0 to 10 (0="not confident", 10="very confident")

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University Frances Payne Bolton School of Nursing, Cleveland, Ohio, United States